CLINICAL TRIAL: NCT06704113
Title: Analgesic Efficacy of Meloxicam Versus Ibuprofen for Pain Control After Third Molar Extraction in Adult Patients: Randomized Clinical Trial
Brief Title: Meloxicam Versus Ibuprofen for Pain Control After Third Molar Exodontia in Adult Patients
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad Austral de Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MelvsIbu
Record Dates: First submitted 2024-07-05; First posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Dental Pain; Sensation Disorders
Keywords: Tooth Extraction; Molar, Third; Meloxicam; Ibuprofen
MeSH Terms: conditions — Toothache; Sensation Disorders | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A control. Ibuprofen (Active Comparator): Ibuprofen 400mg tablets, 1 every 8 hours for 3 days will be administered for post-surgical pain.
  Interventions: Drug: meloxicam 7,5mg
- Group B experimental. Meloxicam (Active Comparator): Meloxicam 7.5mg tablets, 1 every 12 hours for 3 days will be administered for post-surgical pain.
  Interventions: Drug: meloxicam 7,5mg

INTERVENTIONS:
Drug: meloxicam 7,5mg — Comparison of analgesic efficacy of Meloxicam Vs Ibuprofen
  Other Names: ibuprofen 400mg

SUMMARY:
Third molar extraction is a common dental procedure, offently related with pain and swelling. The purpose of this study is to evaluate if Meloxicam has a better effect relieving pain after the extraction than Ibuprofen, one of the most common pain relieving drugs administered after this procedure.

DETAILED DESCRIPTION:
Summary: Third molar extractions are one of the most common procedures in dental practice. However, pain and swelling as postoperative sequelae are inevitable. Depending on the level of pain, which can range from moderate to severe, this symptomatology can be accompanied with pharmacological treatment, thus generating a less traumatic recovery for the patient. It is currently known that non-steroidal anti-inflammatory drugs (NSAIDs) have proven to be effective for the treatment of mild and moderate postoperative pain. Due to the wide variety of NSAIDs, it is important to know how to choose the most effective option when indicating one therapeutic option over another.

Objective: To evaluate the postoperative analgesic effectiveness of meloxicam (7.5 mg) compared to ibuprofen (400 mg) in patients undergoing third molar(s) extraction.

Design: Randomized controlled clinical trial, double-masked, designed according to CONSORT guideline requirements.

ELIGIBILITY:
Inclusion Criteria:

Maxillary or mandibular third molar with semi or fully erupted crown.

Exclusion Criteria:

Patients with Systemic pathologies. Presence of third molar localized infection. Completely included third molar crown. Periodontal compromise. Pregnant or breastfeeding women. Patients with hypersensitivity to NSAIDs. Patients with a history of drug abuse. Patients who had taken any drug in the previous 24 hours. Intervention (exodontia) time longer than 45 minutes.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-12-15 (Estimated); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-01-20 (Estimated)

PRIMARY OUTCOMES:
Meloxicam effectiveness for post-surgical pain control. | 3 days
  A visual analogue scale ranging from 0 points (no pain) to 10 points (intolerable pain) will be used to measure post-exodontic pain, and values will be recorded on a questionnaire.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haffar A, Fillingham YA, Breckenridge L, Gursay D, Lonner JH. Meloxicam versus Celecoxib for Postoperative Analgesia after Total Knee Arthroplasty: Safety, Efficacy and Cost. J Am Acad Orthop Surg Glob Res Rev. 2022 Apr 5;6(4):e22.00032. doi: 10.5435/JAAOSGlobal-D-22-00032. PMID 35389917
- [Background] Iqbal AM, Shetty P. Effect of Submucosal Injection of Tramadol on Postoperative Pain After Third Molar Surgery. J Oral Maxillofac Surg. 2019 Sep;77(9):1752-1759. doi: 10.1016/j.joms.2019.03.029. Epub 2019 Mar 29. PMID 31026419
- [Background] Moore RA, Derry S, Aldington D, Wiffen PJ. Single dose oral analgesics for acute postoperative pain in adults - an overview of Cochrane reviews. Cochrane Database Syst Rev. 2015 Sep 28;2015(9):CD008659. doi: 10.1002/14651858.CD008659.pub3. PMID 26414123
- [Background] Schulz KF, Altman DG, Moher D. CONSORT 2010 statement: Updated guidelines for reporting parallel group randomised trials. J Pharmacol Pharmacother. 2010 Jul;1(2):100-7. doi: 10.4103/0976-500X.72352. No abstract available. PMID 21350618
- [Background] Vallecillo C, Vallecillo-Rivas M, Galvez R, Vallecillo-Capilla M, Olmedo-Gaya MV. ANALGESIC EFFICACY OF TRAMADOL/DEXKETOPROFEN VS IBUPROFEN AFTER IMPACTED LOWER THIRD MOLAR EXTRACTION: A RANDOMIZED CONTROLLED CLINICAL TRIAL. J Evid Based Dent Pract. 2021 Dec;21(4):101618. doi: 10.1016/j.jebdp.2021.101618. Epub 2021 Jul 28. PMID 34922724